CLINICAL TRIAL: NCT01456611
Title: A Double-Blind, Randomized, Placebo-Controlled, Parallel Group, Multi-Site Study to Evaluate the Clinical Equivalence of Diclofenac Sodium 1% Gel (Anchen Pharmaceuticals, Inc.) With Voltaren® Gel (Diclofenac Sodium Topical Gel) 1% (Novartis) in Patients With Osteoarthritis of the Knee
Brief Title: Evaluation of Clinical Endpoints of Two Diclofenac Sodium Gel 1%
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Anchen Pharmaceuticals, Inc (Industry)
Collaborators: Novum Pharmaceutical Research Services (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: DCL-269
Record Dates: First submitted 2011-10-18; First posted 2011-10-21 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Osteo Arthritis of the Knee
MeSH Terms: interventions — Diclofenac

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Diclofenac Sodium Gel (Experimental): Diclofenac sodium Topical Gel 1%
  Interventions: Drug: Diclofenac
- Voltaren (R) Gel (Active Comparator): Voltaren (R) Gel 1%
  Interventions: Drug: Diclofenac
- Placebo (Placebo Comparator): Placebo Topical Gel
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Diclofenac — Diclofenac Sodium Gel 1%
  Arms: Diclofenac Sodium Gel; Voltaren (R) Gel
Drug: Placebo — Placebo Topical Gel
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate the clinical equivalence and safety of the Test formulation of diclofenac sodium topical gel 1% (Anchen Pharmaceuticals, Inc.) compared to the marketed formulation Voltaren® Gel (diclofenac sodium topical gel) 1% (Novartis) in patients with osteoarthritis of the knee.

The efficacy of both the Test and Reference formulations will also be compared to the Placebo gel to determine Superiority.

ELIGIBILITY:
Inclusion Criteria:

1. Ambulatory Male and Non Pregnant Females 35 years and older diagnosed with osteoarthritis (according to the American College of Rheumatology Criteria) in one or both knees.

ACR Criteria includes, Knee Pain and at least 3 of the following:

1. age ≥ 50
2. stiffness lasting < 30 mins
3. bony tenderness
4. crepitus
5. bony enlargement
6. no palpable warmth

2. Symptom onset of > 6 Months prior to Screening for the target knee.

3. If female and of child-bearing potential, prepare to abstain from sexual intercourse or use a reliable method of contraception during the study (e.g., condom + spermicide, IUD, oral, transdermal, injected or implanted hormonal contraceptives).

4. Periarticular knee pain due to osteoarthritis (not bursitis, tendonitis etc) requiring the use of oral or topical treatments (NSAIDS or acetaminophen) for > 15 days in the 30 days prior to Screening.

5. Radiograph of the target knee within the previous year with a Grade 1, 2 or 3 disease based upon the Kellgren-Lawrence disease severity scale.

6. After a 7 day wash out of all pain medication has baseline pain on movement score of ≥ 50mm on a 100-mm Visual Analogue Scale for the target knee.

7. After a 7 day wash out of all pain medication has baseline WOMAC pain sub scale of ≥ 9 on a 5 question, 5 point (0 to 4) Likert scale for the target knee.

8. Willing and able to use only acetaminophen as rescue medication

9. Willing and able to comply with the study requirements.

Exclusion Criteria:

1. Females who are pregnant, breast feeding, or planning a pregnancy
2. Radiograph of the target knee within the previous year with a Grade 4 score on the Kellgren-Lawrence disease severity scale. 24
3. History of osteoarthritis in the contralateral knee requiring medication (OTC or prescription) within 12 months of screening.
4. After a 7 day wash out of all pain medication has baseline pain on movement score of ≥ 20mm on a 100-mm Visual Analogue Scale for the contralateral knee immediately prior to randomization.
5. Known history of secondary osteoarthritis (e.g. congenital, traumatic, gouty arthritis) or rheumatoid arthritis.
6. Known history of other chronic inflammatory diseases, (e.g.,colitis) or fibromyalgia.
7. History of asthma, hypertension, myocardial infarction, thrombotic events, stroke, congestive heart failure, impaired renal function or liver disease.
8. History of coronary artery bypass graft within 6 months of screening.
9. Concomitant acetylsalicylic acid therapy other than a stable low dose used for cardiac prophylaxis (max 162mg daily) taken for at least 3 months prior to enrollment and maintained throughout the duration of the study.
10. Use of warfarin or other anticoagulant therapy within 30 days of screening.
11. Use of ACE inhibitors, cyclosporine, diuretics, lithium or methotrexate, within 30 days of screening or during the study.
12. Known history of gastrointestinal bleeding or peptic ulcer disease.
13. Abnormal screening clinical laboratory evaluations which the Investigator determines are clinically significant.
14. Known allergy to aspirin or NSAIDs.
15. Results from liver function tests that are more than two times the upper limit of the normal range at screening.
16. Any other acute or chronic illness that in the opinion of the investigator could compromise the integrity of study data or place the Patient at risk by participating in the study.
17. Concomitant use of corticosteroids (any formulation) or use within 30 days of study randomization.
18. Receipt of any drug as part of a research study within 30 days prior to screening.
19. Previous participation in this study.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 749 (Actual)
Dates: Start 2011-09; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Mean Change from Baseline in WOMAC Pain Scale | Baseline and Week 4

SECONDARY OUTCOMES:
Superiority of Test and Reference against Placebo in the Mean Change from baseline in the total WOMAC pain score. | Baseline and Week 4
  The superiority of treatment over the placebo will be concluded if the treatment's mean change from baseline in the total WOMAC pain score is statistically significantly greater (p<0.05) than that of the placebo in the ANCOVA based on the treatment and placebo results. The superiority of Test and Reference treatments over the placebo will be evaluated identically in a separate ANCOVA.
  The analyses will be conducted in the mITT population.

CONTACTS AND LOCATIONS:
Locations (57):
- United States (57):
  - Novum Investigator Site, Birmingham, Alabama
  - Novum Investigator Site, Huntsville, Alabama
  - Novum Investigator Site, Chandler, Arizona
  - Novum Investigator Site, Mesa, Arizona
  - Novum Investigator Site, Phoenix, Arizona
  - Novum Investigator Site, Tuscon, Arizona
  - Novum Investigator Site, Little Rock, Arkansas
  - Novum Investigator Site, Anaheim, California
  - Novum Investigator Site, Carmichael, California
  - Novum Investigator Site, Garden Grove, California
  - Novum Investigator Site, Long Beach, California
  - Novum Investigator Site, Sacramento, California
  - Novum Investigator Site, San Diego, California
  - Novum Investigator Site, Stock Bridge, California
  - Novum Investigator Site, Denver, Colorado
  - Novum Investigator Site, Norwalk, Connecticut
  - Novum Investigator Site, Stamford, Connecticut
  - Novum Investigator Site, Adventura, Florida
  - Novum Investigator Site, Bookville, Florida
  - Novum Investigator Site, Bradenton, Florida
  - Novum Investigator Site, Daytona Beach, Florida
  - Novum Investigator Site, Hialeah, Florida
  - Novum Investigator Site, Jupiter, Florida
  - Novum Investigator Site, Miami, Florida
  - Novum Investigator Site, Ormond Beach, Florida
  - Novum Investigator Site, Pinellas Park, Florida
  - Novum Investigator Site, Sarasota, Florida
  - Novum Investigator Site, St. Petersburg, Florida
  - Novum Investigator Site, Tampa, Florida
  - Novum Investigator Site, Marietta, Georgia
  - Novum Investigator Site, Sandy Springs, Georgia
  - Novum Investigator Site, Lexington, Kentucky
  - Novum Investigator Site, New Orleans1, Louisiana
  - Novum Investigator Site, Hollywood, Maryland
  - Novum Investigator Site, Billings, Montana
  - Novum Investigator Site, Henderson, Nevada
  - Novum Investigator Site, Cary, North Carolina
  - Novum Investigator Site, Charlotte, North Carolina
  - Novum Investigator Site, Hickory, North Carolina
  - Novum Investigator Site, High Point, North Carolina
  - Novum Investigator Site, Raleigh, North Carolina
  - Novum Investigator Site, Salisbury, North Carolina
  - Novum Investigator Site, Wilmington, North Carolina
  - Novum Investigator Site, Winston-Salem, North Carolina
  - Novum Investigator Site, Cleveland, Ohio
  - Novum Investigator Site, Columbus, Ohio
  - Novum Investigator Site, Beavercreek, Oklahoma
  - Novum Investigator Site, Norman, Oklahoma
  - Novum Investigator Site, Duncansville, Pennsylvania
  - Novum Investigator Site, Chattanooga, Tennessee
  - Novum Investigator Site, Houston, Texas
  - Novum Investigator Site, Longview, Texas
  - Novum Investigator Site, San Antonio, Texas
  - Novum Investigator Site, Sugar Land, Texas
  - Novum Investigator Site, Charlottesville, Virginia
  - Novum Investigator Site, Midlothian, Virginia
  - Novum Investigator Site, Newport News, Virginia